CLINICAL TRIAL: NCT06625502
Title: Unmute's CARE Framework: A Novel Approach to Strengthen the Therapeutic Alliance and Reduce Treatment Disparities
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FY2024-9189
Record Dates: First submitted 2024-09-24; First posted 2024-10-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Depression Scale Score; Anxiety Symptoms; Functioning, Psychosocial; Working Alliance
Keywords: mental health; therapeutic relationship
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARE framework (Experimental): In this single-arm study, all participants will receive the CARE protocol, which includes a) 3-4 session protocol aimed at cultivating the therapeutic alliance across therapist-patient differences, b) therapist and patient collaboration on a case formulation and treatment plan, c) evidence-based approaches to treating the presenting problem, d) alliance-focused training to address ruptures, and e) cultural case consultation.
  Interventions: Behavioral: Culturally-Affirming Racial Equity Framework

INTERVENTIONS:
Behavioral: Culturally-Affirming Racial Equity Framework — The CARE framework is a process-focused, protocol- based, and modular approach to promote mental health equity. It focuses on cultivating the therapeutic alliance across patient-provider differences in the first 3-4 treatment sessions, the critical window for engaging patients in care. Target processes include transparent communication, client-centeredness, client activation, and an affirming and comprehensive approach to assessment and treatment planning. Case conceptualization and treatment planning is collaborative, and guided by the individual clinician based on evidence-based treatments. The therapist receives ongoing biweekly supervision in Alliance-Focused Training and consultation sessions with a group-specific expert.

SUMMARY:
Aim 1: Expand and adapt the CARE framework to train providers to cultivate a strong early alliance with patients who do not share their background (e.g., mismatched dyads). Aim 2: Establish the feasibility, acceptability, and preliminary effectiveness of the adapted CARE framework in mismatched dyads involving 8 providers and 40 patients receiving 15 sessions of teletherapy.

The goal of this clinical trial is to learn if a new CARE intervention works to improve the cultural fit of psychotherapy for diverse populations, even when the therapist and patient do not share the same cultural background. We will refine and test the intervention with a sample of therapists working with Asian American participants receiving short-term individual psychotherapy delivered online.

The main questions the study aims to answer are:

* Does the CARE framework, adapted for and delivered by therapists specifically trained to work with patients who do not share their background (e.g., mismatched dyads), improve treatment engagement and retention?
* Is the CARE framework associated with a) the development of a positive therapeutic relationship between mismatched patient-therapist dyads and b) significant improvements in participants' presenting problems?

Participants will:

* Receive up to 15 weekly sessions of individual psychotherapy
* Complete different online surveys after every session and on a monthly basis

DETAILED DESCRIPTION:
Despite decades of research exploring approaches to tailoring mental health services to meet the needs of a heterogeneous patient population, significant disparities remain. When patients and providers do not share a similar background, it can result in patients' greater reluctance to engage in treatment, lower satisfaction, and a higher likelihood of dropping out of care, resulting in worsening overall health and contributing to over $153B in excess healthcare costs annually. Two promising approaches to addressing this problem- professional development training to raise provider awareness of the issues, and adapting treatments to specific groups- have failed to reduce treatment disparities. First, studies evaluating the effects of training to enhance providers' ability to tailor services to patient needs find that they tend to focus on abstract concepts, without practical training in skills development. Second, although treatments adapted for specific groups are more effective than unadapted treatments, system constraints (time, cost) limit capacity to train clinicians to deliver multiple adapted treatments to different groups with fidelity. Therefore, a major challenge is how to most feasibly and effectively train our provider workforce to deliver effective mental health care to an increasingly heterogeneous patient population.

Unmute has begun to address this challenge by developing the CARE framework, an innovative process-focused, protocol-based, and modular approach that addresses a preference among many patients for short- term, problem-focused, and individually-tailored treatment to reduce health disparities. Unmute's CARE framework targets the assessment and engagement phase of treatment to reduce dropout, emphasizing skills- training for providers to strengthen the therapeutic alliance, a change mechanism robustly associated with treatment outcome in both telehealth and in-person formats, but more difficult to cultivate across patient-provider differences. Providers receive training in 3 core areas: 1) evidence-informed assessment protocols to facilitate tailoring of treatment, 2) alliance-focused training, an evidence-based approach to repairing breakdowns in the alliance, and 3) consultation with experts in working with specific groups to guide the development of a customized case conceptualization and treatment plan. To date, Unmute's CARE framework has been pilot tested with 10 patients, with 100% returning after the first session, and promising evidence of feasibility and acceptability of core model components. Building on these results, the focus of this Phase I proposal is to train a larger cohort of providers to implement Unmute's CARE framework with patients whose backgrounds differ from their own. We hypothesize that this innovative modular approach to provider training and patient engagement, will increase the feasibility, acceptability, and preliminary effectiveness of providers' efforts to cultivate a strong alliance, reduce dropout rates, and improve treatment engagement and outcome.

Aim 1 will be to expand and adapt the CARE framework to train providers to cultivate a strong early alliance with patients who do not share their background (e.g., mismatched dyads). Guided by pilot data and a community advisory board, we will develop two new training modules: a) a group-specific module, and b) a bridging differences module, to strengthen the patient-provider alliance in mismatched dyads.

Aim 2 will be to establish the feasibility, acceptability, and preliminary effectiveness of the adapted CARE framework in mismatched dyads involving 8 providers and 40 patients receiving 15 sessions of teletherapy. We will collect self-report and observer data for evaluation and refinement as needed.

By combining general and group-specific alliance-building components, Unmute's CARE framework can be adapted for other populations to provide high quality, evidence-based care in an efficient and cost-effective way. Our team is well positioned to execute on this plan; Unmute is cofounded by Colleen Leung, serial entrepreneur and MBA graduate of Babson College, and Dr. Doris Chang, clinical psychologist and expert on culture and mental health and psychotherapy process and outcome in mismatched dyads, with support from the Centers of Alliance Focused Training and New York University's Silver School of Social Work.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants:

1. Individuals 18 years of age or older
2. Physically residing in New York or New Jersey and willing to meet therapist over video platform
3. English-language proficient
4. Seeking telemental health treatment and willing to receive short-term treatment (maximum 15 sessions)
5. Willingness to have sessions videorecorded and complete online assessments
6. Has insurance coverage for therapy sessions or willing to pay for services out-of-pocket ($150/session)

Therapist Participants:

1. Masters' or doctoral level mental health provider licensed to practice in NY or NJ and insured
2. 2+ years of clinical experience post-licensure
3. Training and experience with cognitive behavioral therapy or other evidence-based therapies
4. Interest in improving skills in working across therapist-patient differences
5. Willingness to complete post-session questionnaires, record treatment sessions and attend biweekly AFT sessions for training and research purposes
6. Availability to treat a caseload of 5 Unmute patients during the project period

Exclusion Criteria:

Patient Participants:

1. Patient's symptom presentation is severe beyond what can be effectively managed in a short-term treatment modality via telehealth (e.g., PHQ-9 score greater than 20, they present a risk of harm to self or other, or otherwise require a higher level of care)
2. Patient is involved in another intervention study or currently receiving psychotherapy services from another provider.suicidal ideation or psychotic symptoms
3. Therapist Participants: Licensure violations or enforcement actions as documented at the New York State Office of the Professions https://www.op.nysed.gov/ or New Jersey Division of Consumer Affairs https://www.njconsumeraffairs.gov

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Credibility/Expectancy Questionnaire | Week 4 of treatment
  A brief scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies. Given that Asian American have the lowest rates of mental health service utilization and high dropout rates, we will set conservative success criteria for acceptability, defined as (a) a mean score > 5 (on a 1-9 scale) for the 3 credibility items of the Credibility/Expectancy Questionnaire.
Client Satisfaction Questionnaire-8 (CSQ-8) | At the end of treatment, typically at 15 weeks.
  8-item measures of client satisfaction with services
Retention | Through study completion, approximately 15 weeks.
  We will examine retention outcomes, setting the success criteria at 70% returning after the initial session and 50% retention rate (defined as completing at least 1 follow-up assessment). In general, Asian Americans tend to drop out of therapy at a high rate (as high as 80% in some studies, e.g., Presley & Day, 2019). As a result, we will consider a 50% retention rate to be evidence of 'successful' retention in these racially mismatched therapy dyads.

SECONDARY OUTCOMES:
PHQ-9 | Every 4 weeks through study completion (e.g., week 4, week 8, week 12, week 15) and 3 months after treatment ends.
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
GAD-7 | Every 4 weeks through study completion (e.g., week 4, week 8, week 12, week 15) and 3 months after treatment ends.
  The GAD-7 is a valid and efficient tool for screening for Generalized Anxiety Disorder and assessing its severity in clinical practice and research. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%) and post-traumatic stress disorder (sensitivity 66%, specificity 81%).
Outcome Questionnaire 45.2 (OQ45.2) | Every 4 weeks through study completion (e.g., week 4, week 8, week 12, week 15) and 3 months after treatment ends.
  The Interpersonal Relations (IR) and Social Role (SR) sub scales of the OQ-45.2, a self-report scale designed to track and measure client progress in psychotherapy.
Patient Progress on Goals | Every 4 weeks through study completion (e.g., week 4, week 8, week 12, week 15) and 3 months after treatment ends.
  An idiographic assessment of patient&#39;s self-reported progress on up to 3 treatment goals. 1= Not at all Achieved ---- 9= Completely Achieved

OTHER OUTCOMES:
Session Alliance Inventory | 1 week (after every weekly session)
  A 6-item measures of the working alliance, the key target mechanism of action.
Rupture Resolution Questionnaire | 1 week (after every weekly session)
  Six questions (Muran, Safran, Samstag, & Winston, 2002) aimed at providing a global assessment of rupture and resolution within each session. Participants assess the following on a 5-point Likert Scale: (1) whether there was the perception of any problem or tension in the relationship during the session, (2) to what extent there was a perception of "smoothing over" or "holding back", (3) the extent to which the problem was addressed, (4) the degree to which the problem was resolved, (5) a brief description of the problem, and (6) a brief description of how the the resolution.
Multicultural Orientation | Week 1 (Cultural Comfort) and Week 4 (Cultural Humility, and Cultural Broaching/Missed Opportunities)
  The Multicultural Orientation Framework conceptualizes how therapist and client cultural identities interact in therapy to influence the therapeutic relationship, and includes brief standardized measures of client ratings of Therapist Cultural Comfort, Cultural Humility, and Cultural Broaching/Missed Opportunities.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Unmute Enterprise Inc. [A telehealth company], Chelsea, Massachusetts
  - Virtual/Telehealth, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Only patient and therapist survey data will be considered.Data and metadata will be stored in the NIMH Data Archive (NDA). The data will be made available within 6 months of study completion and will be available for up to 5 years.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available within 6 months of study completion and will be available for up to 5 years.
Access Criteria: Participants will be given the option of consenting to share their survey data for research. For all participants who consent to data sharing, we will not restrict sharing of data. Data and metadata will be stored in the NIMH Data Archive (NDA). We will make available copies of the study protocols, variable list and data collection instruments to facilitate interpretation of the quantitative data.

DOCUMENTS (2):
  • Informed Consent Form: Therapist Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT06625502/ICF_000.pdf
  • Informed Consent Form: Patient Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT06625502/ICF_001.pdf